CLINICAL TRIAL: NCT05694468
Title: The Effects of a Relaxation Intervention on College Students' Social-emotional Competence: A Mixed Methods Approach
Brief Title: The Effects of a Relaxation Intervention on College Students' Social-emotional Competence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Évora (Other)
Responsible Party: Principal Investigator, Andreia Dias Rodrigues, Principal Investigator, University of Évora
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 28122022
Record Dates: First submitted 2022-12-28; First posted 2023-01-23 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Stress
Keywords: social-emotional development; body-oriented intervention; stress; higher education

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Control and Intervention group (Other): In this non-random one-group repeated measures study with a mixed approach (quantitative and qualitative analysis), participants were tested on two occasions 4 weeks apart (baseline measure), and then engaged in the psychomotor relaxation program twice weekly for 8 weeks. Participants were tested again after the intervention program (post-test). The participants took part in a psychomotor relaxation program comprised by two 20-minute sessions per week for 8 weeks, with the whole class, and combined body awareness, muscle tone regulation and breathing exercises.
  Interventions: Other: Psychomotor Relaxation

INTERVENTIONS:
Other: Psychomotor Relaxation — Psychomotor relaxation sessions.

SUMMARY:
Objective: To examine the impact of a psychomotor relaxation program on college students' social-emotional competence, personal and professional development. Participants: Twenty female college students participated. Methods: In this non-random one-group repeated measures study with a mixed approach (quantitative and qualitative analysis), participants were tested on two occasions 4 weeks apart (baseline measure), and then engaged in the psychomotor relaxation program twice weekly for 8 weeks. Participants were tested again after the intervention program (post-test).

DETAILED DESCRIPTION:
This was a non-random one-group repeated measures study with a mixed approach (quantitative and qualitative analysis), where participants served as their own controls.

The investigators examined the chronic effects of the intervention program, collecting the instruments online at week 1 (pretest 1) and week 5 (pretest 2), to establish the baseline measures, and at the end of the 8-week period (post-test). In the post-test evaluation, participants also completed the questionnaire with open-ended questions. Investigators also measured salivary cortisol at the beginning and end of the 1st and the 15th sessions to evaluate the acute effects of the intervention program.

Students participated in a psychomotor relaxation program comprised by two 20-minute sessions per week for 8 weeks, combining body awareness, muscle tone regulation and breathing exercises

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 30 years old
* not having participated in a similar intervention program within the last 6 months
* not have a physical condition that can affect participation in the program
* do not take medication that can influence the studied outcomes.

Exclusion Criteria:

* age under 18 or over 30 years old
* have participated in a similar intervention program within the last 6 months
* have a physical condition that can affect participation in the program
* take medication that can influence the studied outcomes.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2021-06-09 (Actual); Study Completion 2021-06-09 (Actual)

PRIMARY OUTCOMES:
Change in Stress | 1, 4 and 12 weeks.
  Stress was measured through the Portuguese version of the Perceived Stress Scale (PSS-10).
Cortisol levels | 2 days
  Cortisol levels (mcg/dL) were quantified in saliva samples collected at the same time and in the same place where the intervention occurred. Before and after the 1st and 15th session, the samples were collected directly from each participant's mouth.
Change in Affective states | 1, 4 and 12 weeks.
  Affective states were measured through the Portuguese short version of the Profile of Mood States (POMS).
Change in Interoceptive awareness | 1, 4 and 12 weeks.
  Interoceptive awareness was measured through the Portuguese version of the Multidimensional Assessment of Interoceptive Awareness (MAIA).
Change in Psychological wellbeing | 1, 4 and 12 weeks.
  Psychological wellbeing was measured through the Portuguese short version of the Scales of Psychological Wellbeing (EBEP).
Personal and professional development | 1 day (after the intervention program)
  A questionnaire was created to the present study comprising 3 open-ended questions concerning the perception of the students about the influence of the intervention program on their personal development, and the benefits that the intervention program may have in the exercise of their future profession as an early childhood educator.

CONTACTS AND LOCATIONS:
Overall Officials: Andreia D Rodrigues, M, Principal Investigator — PhD student
Locations (1):
- Andreia Dias Rodrigues, Evora, Portugal

IPD SHARING:
Plan to Share IPD: No